CLINICAL TRIAL: NCT01234662
Title: Combined Spinal Epidural Anesthesia (CSE) vs Spinal Anesthesia for Elective Cesarean Sections. Influence of Surgical Regional Anesthesia on Postoperative Pain
Brief Title: Influence of Surgical Regional Anesthesia on Postoperative Pain
Acronym: CESAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Christian von Heymann, M.D., Prof. Dr. med. Christian von Heymann, Department of Anesthesiology and Intensive Care Medicine, CVK/CCM, Charite University, Berlin, Germany., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CESAR
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Elective Cesarean Section
Keywords: Elective cesarean sections; Postoperative pain level; Spinal anesthesia; Combined spinal epidural anesthesia; Epidural catheter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Active Comparator): Spinal anesthesia + intrathecal opioid bolus (SPA)
  Interventions: Procedure: SPA
- Group 2 (Active Comparator): CSE + epidural opioid bolus (CSE)
  Interventions: Procedure: CSE
- Group 3 (Experimental): CSE + continuous epidural patient controlled analgesia using an epidural catheter for 24 hrs (CSEPCEA)
  Interventions: Procedure: CSEPCEA

INTERVENTIONS:
Procedure: SPA — Spinal anesthesia and opioids
  Arms: Group 1
Procedure: CSE — CSE and epidural opioids
  Arms: Group 2
Procedure: CSEPCEA — CSE and continuous epidural patient controlled analgesia using an epidural catheter for 24 hrs
  Arms: Group 3

SUMMARY:
To compare three Types of anesthetic techniques (Spinal anesthesia, Combined spinal epidural anesthesia, Combined spinal epidural anesthesia with indwelling catheter for 24 hrs) on pain after elective cesarean section.

DETAILED DESCRIPTION:
Regional analgesia is the most effective way of providing analgesia during labor and delivery. By using a combination of local anesthetics and opioids, it is often possible to avoid motor block. Spinal anesthesia is suitable for most elective cesarean sections. Epidural anesthesia and in particular catheter based epidural anesthesia allow a gradual extension of anesthesia and are suitable for prolonged treatment of postoperative pain.

It is unclear which anesthetic technique provides better pain relief after cesarean section.

This prospective, randomized study compares the effectiveness of three types of regional anesthetic techniques (Spinal anesthesia, Combined spinal epidural anesthesia, Combined spinal epidural anesthesia with indwelling catheter for 24 hrs) on pain after elective cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged greater than or equal to 18 years
* Patients without severe illnesses (American Society of Anaesthesiologists [ASA] grade II-III)
* Patients for elective cesarean sections
* Informing patients about risks and complications of anesthesia until 24 hrs before operation

Exclusion Criteria:

* Lacking willingness to regional procedures
* No offered patient information and written informed consent
* Persons without the capacity to consent
* Unability of German language use
* Preterm delivery < 28 weeks of pregnancy
* Chronic pain or chronic analgesic intake in medical history
* Alcohol, dope and medication abuse
* Psychiatric disease in medical history
* Baby death after delivery
* Anxiolytic medication
* Allergy to local anaesthetics
* History of bleeding tendency
* Eclampsia and HELLP syndrome
* Elective section out work routine time
* Participation in another clinical trial during the trial, one month before screening and three months after screening

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-04 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain levels during movement (cough) | At nine hours after the end of surgery (closure time)
  Patient self-assessed postoperative pain levels during movement (cough) using an unmarked zero to one hundred mm visual analog scale (VAS)

SECONDARY OUTCOMES:
Postoperative pain levels during rest | At nine hours after the end of surgery (closure time)
  Patient self-assessed postoperative pain levels during rest using an unmarked zero to one hundred mm visual analog scale (VAS)
Postoperative pain levels during rest and movement | At zero (injection), one, two, six, nine, twenty four, fourty eight hours after the end of surgery (closure time)
  Patient self-assessed postoperative pain levels during rest and movement using an unmarked zero to one hundred mm visual analog scale (VAS)
Change of type of anesthesia when regional anesthesia fails | During the operation
Level of anesthesia during the operation | During the operation
Incidence of hypotensions during the operation | During the operation
Sedation level (Ramsay-Score) | Postoperative course
Capability for mobilisation and time to first mobilisation | Postoperative course
Incidence of adverse reactions (PONV, headache and backpain, urinary retention) | Postoperative course
Satisfaction with pain management | Postoperative course
Co-analgesics | In the 48-hour postoperative sample period
  Co-analgesic consumption

CONTACTS AND LOCATIONS:
Overall Officials: Christian von Heymann, MD Prof., Study Director — Department of Anesthesiology and Intensive Care Medicine, Campus Virchow Klinikum
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Campus Virchow Klinikum, Campus Charité Mitte, Charite University, Berlin, Berlin, State of Berlin, Germany